CLINICAL TRIAL: NCT04034355
Title: A Phase 3, Double-blind, Multicenter, Placebo-controlled Study of PledOx Used on Top of Modified FOLFOX6 (5-FU/FA and Oxaliplatin) to Prevent Chemotherapy Induced Peripheral Neuropathy (CIPN) in the Adjuvant Treatment of Patients With Stage III or High-risk Stage II Colorectal Cancer
Brief Title: Preventive Treatment of OxaLiplatin Induced peripherAl neuRopathy in Adjuvant Colorectal Cancer
Acronym: POLAR-A
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: On 01 March 2020, the Sponsor decided to place recruitment and dosing of patients on hold following interactions with the French regulatory authority, ANSM and the US clinical hold of another study (POLAR-M).
Sponsor: Egetis Therapeutics (Industry)
Collaborators: Solasia Pharma K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PP06489; 2017-004707-43 (EudraCT Number)
Record Dates: First submitted 2019-05-14; First posted 2019-07-26 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer; Chemotherapy-induced Peripheral Neuropathy
Keywords: colorectal cancer; cancer; peripheral neuropathy; neuropathy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Peripheral Nervous System Diseases | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Intervention Model Description: Patients with colorectal cancer (CRC), who are indicated for adjuvant modified FOLFOX6 (mFOLFOX6) chemotherapy for up to 6 months, will be randomized in a 1:1 ratio to 1 of 2 treatment arms:
  * Arm A: PledOx (5 µmol/kg) + mFOLFOX6 chemotherapy
  * Arm B: Placebo + mFOLFOX6 chemotherapy
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PledOx (5 µmol/kg) (Experimental): Calmangafodipir 5 µmol/kg
  Interventions: Drug: Calmangafodipir (5 µmol/kg)
- Placebo (Placebo Comparator): 0.9% sodium chloride in 20 mL vials
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Calmangafodipir (5 µmol/kg) — PledOx will be given to patients as an i.v. infusion, on top of mFOLFOX6 chemotherapy. PledOx is a solution in 20 mL single dose glass vials.
  Other Names: PledOx
  Arms: PledOx (5 µmol/kg)
Other: Placebo — Placebo will be administered via the same route as PledOx (i.v. infusion). Placebo is a solution in 20 mL single dose glass vials.
  Arms: Placebo

SUMMARY:
This study is to evaluate PledOx for prevention of chronic chemotherapy induced peripheral neuropathy induced by oxaliplatin in patients with Stage III or high-risk Stage II colorectal cancer (CRC).

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, double-blind, placebo-controlled study with PledOx for prevention of chronic CIPN induced by oxaliplatin in patients with Stage III or high-risk Stage II colorectal cancer (CRC).

Patients with CRC, who are indicated for adjuvant modified FOLFOX6 (mFOLFOX6) chemotherapy for up to 6 months, will be randomized in a 1:1 ratio to 1 of 2 treatment arms:

* Arm A: PledOx (5 µmol/kg) + mFOLFOX6 chemotherapy
* Arm B: Placebo + mFOLFOX6 chemotherapy

Before March 2nd., 2020, the investigational medicinal product (IMP; i.e. PledOx or placebo) was administered by an intravenous (i.v.) infusion on the first day of each chemotherapy cycle. IMP was not to be administered if mFOLFOX6 was not given to the patient.

If a patient later discontinues oxaliplatin, treatment with 5-FU/folinate and IMP may be continued.

As of March 2nd., all patients have to stop IMP but may continue mFOLFOX6.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form before any study related assessments and willing to follow all study procedures.
2. Male or female aged ≥18 years.
3. Pathologically confirmed adenocarcinoma of the colon or rectum including: Stage III carcinoma (any T N1,2 M0) or Stage II carcinoma (T3,4 N0 M0).
4. The patient has undergone curative (R0) surgical resection performed within 12 weeks prior to randomization
5. The patient has a postsurgical carcinoembryonic antigen (CEA) level ≤1.5 x upper limit of normal (ULN, in current smokers, CEA level ≤2.0 x ULN is allowed).
6. No prior anti-cancer therapy for CRC except radiotherapy or concomitant chemo-radiotherapy using a fluoropyrimidine alone for locoregional rectal cancer.
7. Patient indicated for up to 6 months of oxaliplatin-based chemotherapy and without pathological findings of a neurologic exam performed prior to oxaliplatin treatment according to local practice.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Adequate hematological parameters: hemoglobin ≥100 g/L, absolute neutrophil count ≥1.5 x 109 /L, platelets ≥100 x 109 /L.
10. Adequate renal function: creatinine clearance >50 cc/min using the Cockcroft and Gault formula or measured.
11. Adequate hepatic function: total bilirubin ≤1.5 x ULN (except in the case of known Gilbert's syndrome); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x ULN.
12. Baseline blood manganese (Mn) level <2.0 x ULN.
13. For patients with a history of diabetes mellitus, HbA1c ≤7%.
14. Negative pregnancy test for women of child-bearing potential (WOCBP).
15. For men and WOCBP, use of adequate contraception (oral contraceptives, intrauterine device or surgically sterile) while on study drug and for at least 6 months after completion of study therapy.

Exclusion Criteria:

1. Any evidence of metastatic disease.
2. Any unresolved toxicity by National Cancer Institute-Common Terminology Criteria for Adverse Events Version (NCI-CTCAE) v.4.03 >Grade 1 from previous anti-cancer therapy (including radiotherapy), except alopecia.
3. Any grade of neuropathy from any cause.
4. Any evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, cardiac, unresolved bowel obstruction, hepatic or renal disease).
5. Chronic infection or uncontrolled serious illness causing immunodeficiency. Patients with known history of chronic hepatitis B can be enrolled if they are asymptomatic and an acute and active HBV infection can be excluded.
6. Any history of seizures.
7. A surgical incision that is not healed.
8. Known hypersensitivity to any of the components of mFOLFOX6 and, if applicable, therapies to be used in conjunction with the chemotherapy regimen or any of the excipients of these products.
9. History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within 5 years, unless the patient has been disease free for that other malignancy for at least 2 years.
10. Known dihydropyrimidine dehydrogenase deficiency.
11. Pre-existing neurodegenerative disease (e.g., Parkinson's, Alzheimer's, Huntington's) or neuromuscular disorder (e.g., multiple sclerosis, amyotrophic lateral sclerosis, polio, hereditary neuromuscular disease).
12. Major psychiatric disorder (major depression, psychosis), alcohol and/or drug abuse.
13. Patients with a history of second or third degree atrioventricular block or a family heredity.
14. A history of a genetic or familial neuropathy.
15. Treatment with any investigational drug within 30 days prior to randomization.
16. Pregnancy, lactation or reluctance to using contraception.
17. Any other condition that, in the opinion of the Investigator, places the patient at undue risk.
18. Previous exposure to mangafodipir or calmangafodipir.
19. Welders, mine workers or other workers in occupations (current or past) where high Mn exposure is likely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Carlsson, MD, Study Director — Chief Medical Officer
Locations (65):
- Belgium (8):
  - Onze-Lieve-Vrouwziekenuis Aalst, Aalst
  - Imelda GI Clinical Research Center, Bonheiden
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Gent, Ghent
  - CHU Liège, Liège
  - AZ Sint Maarten, Mechelen
  - AZ Delta, Roeselare
  - CHU UCL Namur - Site Godinne, Yvoir
- Czechia (5):
  - Nemocnice Benesov, Benešov
  - Nemocnice Horovice, Hořovice
  - Nemocnice Na Pleši, Nová Ves Pod Plesi
  - General University Hospital, Prague
  - Onkologická Klinika 1. Lf Uk A Tn, Prague
- France (9):
  - CHRU de Brest - Hôpital Morvan, Brest
  - Clinique Pasteur-Lanroze, Brest
  - Centre Hospitalier Départemental de Vendée - Unité de recherche clinique, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Hôpital Edouard Herriot - HCL, Lyon
  - Hôpital Nord Franche-Comté Site du Mittan, Montbéliard
  - CHU Nice L'Archet 2, Nice
  - Clinique Ste Anne, Strasbourg
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Germany (5):
  - Hämatolgisch-onkologische Praxis Augsburg, Augsburg
  - Onkozentrum Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Onkodok GmbH / Onkologische Schwerpunktpraxis, Gütersloh
  - Klinikum Neuperlach, München
- Italy (8):
  - Oncologia Istituti Ospitalieri, Cremona
  - Irccs Irst, Meldola - FC
  - Hospital San Gerardo, Monza
  - Istituto Nazionale Tumori, Napoli
  - IRCCS Policlinico San Matteo, Pavia
  - Ospedale degli infermi, Ponderano
  - IRCCS azienda Ospedaliera S Maria Nuova, Reggio Emilia
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Japan (11):
  - Fukuoka University Hospital, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - St. Marianna University School of Medicine Hospital, Kawasaki
  - Aichi Cancer Center Hospital, Nagoya
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Osaka University Hospital, Osaka
  - Sapporo Medical University Hospital, Sapporo
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Fujita Health University Hospital, Toyoake
- South Korea (6):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Dong-A University Hospital, Busan
  - Chonnam National University Hwasun Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (8):
  - Granvia de L´Hospitalet 199-203, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Vall d'hebron university hospital, Barcelona
  - Centro Integral Oncologico, Madrid
  - H.G.U.Gregorio Marañón, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Univ Virgen Macarena, Seville
  - Hospital Quironsalud Valencia, Valencia
- KMUH: Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan
- United Kingdom (4):
  - Mid Essex Hospital Services NHS Trust - Broomfield Hospital, Chelmsford
  - North Tyneside General Hospital, North Shields
  - Mount Vernon Cancer Centr, Northwood
  - The Royal Marsden Hospital (Surrey), Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfeiffer P, Lustberg M, Nasstrom J, Carlsson S, Persson A, Nagahama F, Cavaletti G, Glimelius B, Muro K. Calmangafodipir for Prevention of Oxaliplatin-Induced Peripheral Neuropathy: Two Placebo-Controlled, Randomized Phase 3 Studies (POLAR-A/POLAR-M). JNCI Cancer Spectr. 2022 Nov 1;6(6):pkac075. doi: 10.1093/jncics/pkac075. PMID 36308441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the EU and Asia between 7 January 2019 and 1 March 2020. The Sponsor placed recruitment/dosing in the POLAR program on hold following interactions with the French regulatory authority and the US clinical hold of study POLAR-M on 23 January 2020. As of 2 March 2020, no more patients were enrolled or IMP administered. Enrolled patients were followed until the data cut-off date of 31 August 2020 and these patients have been assigned as "completed" in the disposition.
Pre-assignment Details: 371 patients were screened in the 28 days before the start of treatment, 301 were randomised and 297 were treated.
Period: Overall Study
Arm/Group | PledOx (5 µmol/kg) | Placebo
Started | 151 | 150
Treated | 147 | 150
Completed | 117 | 115
Not Completed | 34 | 35
Not completed — Study terminated by Sponsor | 10 | 17
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Site terminated by Sponsor | 4 | 5
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 1
Not completed — Not reported | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Progressive disease | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisting of all randomized patients who received at least one dose of IMP. Patients were analyzed according to the study treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | PledOx (5 µmol/kg) | Placebo | Total
Number analyzed (Participants) | 147 | 150 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (10.4) | 62.4 (10.2) | 62.9 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 61 | 130
  Male | 78 | 89 | 167
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 43 | 43 | 86
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 87 | 93 | 180
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 14 | 29
Body Mass Index [Median (Full Range); unit: kg/m^2] | 24.20 [16.9 to 38.9] | 23.60 [16.8 to 49.7] | 24.20 [16.8 to 49.7]
ECOG performance status [Count of Participants; unit: Participants] — The ECOG performance scale is a six point functional scale (0 to 5) rating the extent of effect on daily living with higher scores representing a worse outcome. A score 0 represents "fully active, able to carry on all pre-disease performance without restriction" and a score 1 represents "restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work".
  Participants
    0 | 118 | 122 | 240
    1 | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Moderate or Severe Chronic Chemotherapy Induced Peripheral Neuropathy (CIPN)
Description: Percentage of patients (with moderate or severe chronic CIPN) scoring 3 or 4 in at least 1 of the first 4 items of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-13-item subscale (FACT/GOG-NTX-13; i.e., FACT/GOG-NTX-4) 9 months after the first dose of IMP (i.e. PledOx or placebo administered on Day 1, Cycle 1 of mFOLFOX6 chemotherapy). The FACT/GOG-13 questionnaire includes 13 items that measure the severity and impact of symptoms of neurotoxicity over the past 7 days. Patients rate each item as 0 ("not at all"), 1 (" a little bit"), 2 ("somewhat"), 3 ("quite a bit") or 4 ("very much"). These 13 items are summed to create a total score, ranging from 0 to 52, with a higher score representing a worse outcome. The FACT/GOG-NTX-4 is a 4 item subscale targeting numbness, tingling or discomfort in hands and/or feet.
Time Frame: 9 months
Population: Modified ITT (mITT) analysis set including patients that fulfilled at least one of the following criteria:
  * the patient was randomized prior to 1 Dec 2019 (i.e. the patient was eligible for at least 3 months of IMP) and had at least one post-baseline assessment for efficacy, or
  * the 3 month Assessment Visit occurred prior to 1 Mar 2020, or
  * the patient received the 6th cycle of IMP after 1 Mar 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 120 | 119
Participants | 68 | 46
Statistical Analysis 1: Comparison: PledOx (5 µmol/kg) vs Placebo; Test type: Superiority; p = 0.0280, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.5210, 95% CI 2-sided [1.0462 to 2.2113]

2. Secondary Outcome: Mild, Moderate or Severe Chronic Chemotherapy Induced Peripheral Neuropathy
Description: Percentage of patients (with mild, moderate or severe chronic CIPN) scoring 2, 3 or 4 in at least 1 of the first 4 items of the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity-13-item subscale (FACT/GOG-NTX-13; i.e., FACT/GOG-NTX-4) 9 months after the first dose of IMP (i.e. PledOx or placebo administered on Day 1, Cycle 1 of mFOLFOX6 chemotherapy). The FACT/GOG-13 questionnaire includes 13 items that measure the severity and impact of symptoms of neurotoxicity over the past 7 days. Patients rate each item as 0 ("not at all"), 1 (" a little bit"), 2 ("somewhat"), 3 ("quite a bit") or 4 ("very much"). These 13 items are summed to create a total score, ranging from 0 to 52, with a higher score representing a worse outcome. The FACT/GOG-NTX-4 is a 4 item subscale targeting numbness, tingling or discomfort in hands and/or feet.
Time Frame: 9 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 120 | 119
Participants | 89 | 74

3. Secondary Outcome: Sensitivity to Touching Cold Items
Description: Mean change from baseline in sensitivity to touching cold items on Day 2, Cycle 4 (cycle is 14 days) of mFOLFOX6 chemotherapy, as assessed by the Cold Sensitivity questionnaire. Cold sensitivity was rated 0 (not at all) to 10 (as bad as you can imagine).
Time Frame: Baseline and 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 120 | 126
Scores on a scale | 4.38 [3.85 to 4.92] | 4.08 [3.55 to 4.61]

4. Secondary Outcome: Cumulative Dose of Oxaliplatin During Chemotherapy
Description: Mean cumulative dose of oxaliplatin administered per patient during mFOLFOX6 chemotherapy, 9 months after the first dose of Investigational Medicinal Product
Time Frame: 9 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/m^2
Arm/Group | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 138 | 140
mg/m^2 | 747.3 [705.5 to 789.2] | 755.0 [713.3 to 796.6]

5. Secondary Outcome: Vibration Sensitivity on the Lateral Malleolus
Description: Mean change from baseline in vibration sense, on the lateral malleolus (left and right), using a graduated tuning fork, at 9 months after the first dose of Investigational Medicinal Product. When the tuning fork was struck against the ball of the thumb, the base of the tuning fork was placed over the appropriate bony surface (i.e. lateral malleolus left and right) and the patient was asked to indicate the moment when the vibration was no longer detected. The intensity at which the patient no longer detected the vibration is reported on a scale of 0 (minimum score, representing the maximum vibration amplitude) to 8 (maximum score, representing the minimum vibration amplitude)
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 108 | 107
Scores on a scale | -1.38 (1.61) | -1.43 (1.84)

6. Secondary Outcome: Worst Pain in Hands or Feet
Description: Mean change from baseline in worst pain in hands or feet in the past week, using a numerical rating scale (Numeric Rating Scale; Scale range of 0-10;0 = no pain, 10= pain as bad as you can imagine), at 9 months after the first dose of Investigational Medicinal Product
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 114 | 118
Scores on a scale | 2.55 [1.97 to 3.14] | 2.16 [1.58 to 2.74]

7. Secondary Outcome: Functional Impairment (in the Non-dominant Hand)
Description: Mean change from baseline in the time to complete the grooved Pegboard with the non-dominant hand, at 9 months after the first dose of Investigational Medicinal Product
Time Frame: Baseline and 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 104 | 107
seconds | 16.23 (48.91) | -0.39 (42.58)

8. Secondary Outcome: Patients With Disease Free Survival
Description: Patients with disease free survival.
Time Frame: Analysis was planned at 24 months but performed based on available data at cut-off 31 August 2020 as the study was terminated early by the Sponsor
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | PledOx (5 µmol/kg) | Placebo
Number analyzed (Participants) | 147 | 150
participants | 7 | 15

ADVERSE EVENTS:
Time Frame: From screening until 30 days after the end of treatment visit which occurred after up to 6 months of treatment
Arm/Group | PledOx (5 µmol/kg) | Placebo
All-Cause Mortality (participants affected / at risk) | 1/147 | 1/150
Serious Adverse Events (participants affected / at risk) | 20/147 | 20/150
Other Adverse Events (participants affected / at risk) | 146/147 | 146/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PledOx (5 µmol/kg) (N=147) | Placebo (N=150)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Administration site cellulitis (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Infusion related reaction (Immune system disorders) | 3 (5) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal stoma complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetitie (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Device extrusion (Product Issues) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PledOx (5 µmol/kg) (N=147) | Placebo (N=150)
Anaemia (Blood and lymphatic system disorders) | 17 (24) | 17 (20)
Leukopenia (Blood and lymphatic system disorders) | 18 (34) | 19 (40)
Neutropenia (Blood and lymphatic system disorders) | 62 (144) | 68 (203)
Thrombocytopenia (Blood and lymphatic system disorders) | 46 (69) | 58 (134)
Abdominal pain (Gastrointestinal disorders) | 13 (18) | 14 (18)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9) | 15 (21)
Constipation (Gastrointestinal disorders) | 30 (38) | 25 (39)
Diarrhoea (Gastrointestinal disorders) | 59 (120) | 56 (90)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 11 (13)
Nausea (Gastrointestinal disorders) | 88 (193) | 69 (155)
Stomatitis (Gastrointestinal disorders) | 50 (67) | 31 (37)
Vomiting (Gastrointestinal disorders) | 27 (33) | 27 (34)
Asthenia (General disorders) | 32 (87) | 36 (73)
Fatigue (General disorders) | 39 (61) | 36 (78)
Malaise (General disorders) | 8 (23) | 7 (9)
Pyrexia (General disorders) | 10 (13) | 13 (18)
Infusion related reaction (Immune system disorders) | 8 (9) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (8) | 7 (7)
Alanine aminotransferase increased (Investigations) | 11 (18) | 17 (26)
Aspartate aminotransferase increased (Investigations) | 11 (19) | 15 (23)
Decreased appetite (Metabolism and nutrition disorders) | 42 (66) | 37 (62)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 11 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (12) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 5 (8) | 8 (12)
Dizziness (Nervous system disorders) | 11 (14) | 4 (4)
Dysaesthesia (Nervous system disorders) | 7 (15) | 13 (22)
Dysgeusia (Nervous system disorders) | 35 (43) | 34 (47)
Headache (Nervous system disorders) | 12 (14) | 13 (18)
Neuropathy peripheral (Nervous system disorders) | 67 (187) | 73 (217)
Paraesthesia (Nervous system disorders) | 30 (82) | 33 (98)
Peripheral sensory neuropathy (Nervous system disorders) | 49 (132) | 39 (129)
Insomnia (Psychiatric disorders) | 8 (8) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 12 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 23 (25) | 18 (19)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 (29) | 15 (21)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5)
Hypertension (Vascular disorders) | 11 (16) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04034355/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT04034355/SAP_001.pdf